CLINICAL TRIAL: NCT05355168
Title: Neoadjuvant Chemoradiotherapy Combined With Camrelizumab and Nimotuzumab for Initially Inoperable Patients With Locally Advanced Esophageal Squamous Cell Carcinoma: A Prospective, One-arm, Phase II Study (NCRCN)
Brief Title: Neoadjuvant CRT Combined With Camrelizumab and Nimotuzumab for Initially Inoperable Patients With Esophageal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Dong Qian, Professor, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-ky238
Record Dates: First submitted 2022-04-16; First posted 2022-05-02 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Toxicity, Drug
Keywords: Esophageal squamous cell carcinoma; neoadjuvant chemoradiotherapy; nimotuzumab; camrelizumab
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Esophageal Squamous Cell Carcinoma | interventions — camrelizumab

STUDY DESIGN:
Intervention Model Description: To enroll 35 initially inoperable patients with locally advanced esophageal squamous cell carcinoma to receive neoadjuvant chemoradiotherapy combined with Camrelizumab and Nimotuzumab followed by surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant treatment (Experimental): Neoadjuvant chemoradiotherapy combined with Camrelizumab and Nimotuzumab
  Interventions: Drug: neoadjuvant chemoradiotherapy combined with Camrelizumab and Nimotuzumab followed by surgery

INTERVENTIONS:
Drug: neoadjuvant chemoradiotherapy combined with Camrelizumab and Nimotuzumab followed by surgery — neoadjuvant chemoradiotherapy combined with Camrelizumab and Nimotuzumab followed by surgery

SUMMARY:
Neoadjuvant chemoradiotherapy followed by surgery has been the standard modality for locally advance esophageal carcinoma. According to CROSS study, the pathological complete remission rate achieved by paclitaxel and carboplatin with 41.4 Gy/23f was 49% for esophageal squamous cell carcinoma. But the 10-year overall survival rate was only 38%. How to increase the overall survival of esophageal carcinoma is a pivotal task. Both of Camrelizumab and Nimotuzumab have been demonstrated to be efficacious in the neoadjuvant treatment for esophageal squamous cell carcinoma in some small sample-size trials. Therefore, this trial is designed to combine adjuvant chemoradiotherapy with Camrelizumab and Nimotuzumab for resectable & potentially resectable locally advanced esophageal squamous cell carcinoma and explore the safety and primary efficacy of such combination.

DETAILED DESCRIPTION:
Trial Title Neoadjuvant chemoradiotherapy combined with Camrelizumab and Nimotuzumab for initially inoperable patients with locally advanced esophageal squamous cell carcinoma: A Prospective, One-arm, Phase II study (NCRCN) Trial Objective To explore the safety and primary efficacy of neoadjuvant chemoradiotherapy combined with Camrelizumab and Nimotuzumab for initially inoperable patients with locally advanced esophageal squamous cell carcinoma.

Trial Design: To enroll 35 patients with initially inoperable patients with locally advanced esophageal squamous cell carcinoma to receive neoadjuvant chemoradiotherapy combined with Camrelizumab and Nimotuzumab followed by surgery.

Staging Examination before Adjuvant Treatment: a. ECOG scoring. b. PET-CT, Upper GI endoscopy & endoscopic ultrasound and barium swallow (preferred), or chest contrast CT, abdominal ultrasonography, bone scan, Upper GI endoscopy & endoscopic ultrasound and barium swallow. c. Bronchoscopy for patients with suspicious invasion into trachea or bronchus. d. Pulmonary function test.

Adjuvant chemoradiotherapy Radiotherapy CT Simulation: CT with intravenous contrast is recommended for simulation. Scan thickness should be less than 5 mm from lower margin of mandibular to lower margin of L2. Thermal mask is recommended.

Delineation of Targets: Involved field irradiation is the general principle. Gross Tumor Volume (GTV) is the primary esophageal tumor and the metastatic lymph node. The Clinical Target Volume (CTV) provided a proximal and distal margin of 3 cm and a 0.8 cm radial margin around the primary esophageal tumor and a proximal and distal margin of 1 cm and a 0.8 cm radial margin around the metastatic lymph nodes. The Planning Target Volume (PTV) was defined as an 8-mm margin of the CTV for tumor motion and set-up variations.

Prescription Dose: 41.4 Gy/23f to PTV. Dosimetric Limitation of Organ at Risk: 95% prescription dose should cover 100% PTV and 95% PTV should receive 100% prescription dose. Total Lung: V20<25%, Dmean<13Gy, V5<50%. Spinal Cord: Dmax<45Gy. Heart: V30<40%, Dmean<25Gy.

Treatment Implementation: Radiotherapy is implemented every day. Cone-beam CT should utilized every week to minimize set-up error.

Chemotherapy nab-paclitaxel 50mg/m2+Carboplatin AUC=2 qw×5c, Nimotuzumab 200mg q3w×2c, Camrelizumab 200mg q3w×2c.

Restaging Examination before Surgery: a. ECOG scoring. b. PET-CT and barium swallow (preferred), or chest contrast CT, abdominal ultrasonography, bone scan and barium swallow. c. Pulmonary function test.

Restaging is aiming to exclude patients with disease progression after neoadjuvant treatment.

Surgery Surgery is scheduled for 4 to 6 weeks after completion of adjuvant treatment. McKeown or Ivor-Lewis esophagectomy, including two-field lymphadenectomy with total mediastinal lymph node dissection, is performed. The dissection of left and right recurrent laryngeal nerve nodes is mandatory.

Follow-up: Patients should be follow-up every three months right after the completion of surgery to 2 years after surgery. Then follow-up every half year is allowed to 5 years after surgery. After 5 years, follow-up every year is appropriate. In follow-up, chest contrast CT and abdominal ultrasonography should be implemented. Endoscopy should be undertaken every year for all patients.

Primary Endpoint: 1-year progression free survival (PFS) rate. Secondary Endpoint: Pathological complete remission rate and major pathological remission rate (CAP Cancer Protocol for Esophageal Carcinoma). Surgical conversion rate, Rate of adverse events (CTCAE V4.0), 2-year progression free survival (PFS) rate.1-year, 2-year overall survival rates (OS) .

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old;
* Eastern Cooperative Oncology Group (ECOG) 0-1;
* Esophageal squamous cell carcinoma;
* cT2-4aN0-3M0-1a (AJCC 8th) confirmed by radiological examination;
* Initially inoperable at initial diagnosis confirmed by thoracic surgeons;
* No esophageal hemorrhage and no esophageal fistula at initial diagnosis;
* Treatment naive;
* No contraindications for adjuvant chemoradiotherapy, camrelizumab and nimotuzumab;
* Signature of inform consent.

Exclusion Criteria:

* younger than 18 years old or older than 75 years old;
* ECOG>1;
* Esophageal adenocarcinoma, small-cell cancer and other pathological types;
* Presence of esophageal hemorrhage and esophageal fistula at initial diagnosis;
* Previous treatment of chemotherapy, radiotherapy, immune therapy and other treatment;
* Contraindications for chemoradiotherapy, camrelizumab and nimotuzumab;
* No signature of inform consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
1-year progression free survival (PFS) rate | 0 month post neoadjuvant treatment
  1-year progression free survival (PFS) rate

SECONDARY OUTCOMES:
Rate of adverse events | 1 to 2years
  Rate of adverse events (CTCAE V4.0)
Pathological complete remission rate | 0 month post surgery
  Pathological complete remission rate (CAP Cancer Protocol for Esophageal Carcinoma)
1-, 2-year overall survival rate . | 1 to 2years
  1-, 2-year overall survival rate .
Major pathological remission rate | 0 month post surgery
  Major pathological remission rate (CAP Cancer Protocol for Esophageal Carcinoma)
surgical conversion rate | 0 month post neoadjuvant
  surgical conversion rate

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provicial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He Y, Liu H, Li X, Wang J, Wu H, Zhou H, Wang X, Cheng J, Ma J, Mei X, Tian J, Qian D. Neoadjuvant chemoradiation with camrelizumab and nimotuzumab for initially inoperable esophageal squamous cell carcinoma: A single-arm phase 2 trial. Eur J Cancer. 2025 Oct 1;228:115717. doi: 10.1016/j.ejca.2025.115717. Epub 2025 Aug 15. PMID 40834785